CLINICAL TRIAL: NCT05482165
Title: Optimizing Intervention Effects in Children and Adolescents in Ningbo City
Brief Title: Optimizing Intervention Effects in Children and Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-R168
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The students of this group will receive multi-faceted intervention activities toward weight management.
  Interventions: Behavioral: Multi-faceted health promotion programme
- Usual practice group (No Intervention): The students of this group will receive regular health education.

INTERVENTIONS:
Behavioral: Multi-faceted health promotion programme — This intervention programme will target the influencing factors of childhood obesity to influence the knowledge, attitude and behaviours of school children. Students in the intervention group will receive the following interventions:
  * Develop and implement school policies related to weight loss
  * Distribute health education materials on diet and exercise to students
  * Carry out student health education courses
  Arms: Intervention group

SUMMARY:
Childhood obesity is a significant public health concern worldwide. In China, childhood obesity has dramatically increased as the economy has grown quickly over the past decades. Effective strategies to reduce childhood obesity prevalence may help to prevent related chronic diseases in the whole population in the long term.

This study aimed (1)to assess the effectiveness of the intervention compared with the usual practice in preventing childhood overweight and obesity; (2) to determine the sustainability of the intervention in preventing overweight and obesity; and (3) to evaluate the process and health economics of the intervention.

The project will be carried out in six primary schools in Ningbo City, Zhejiang Province , those schools are randomly divided into two groups: the intervention group and the usual practice group. The participants of the study were students in the third grade of primary school, and the intervention will last for one academic year. This intervention programme will target the influencing factors of childhood obesity at both individual (student-focused activities) and environmental levels (a supportive family and school environment), with the intent to influence the knowledge, attitude and behaviours of school children.

ELIGIBILITY:
Inclusion Criteria:

* Parents agree and support their children's weight loss, and students and parents have informed consent;
* Students in third grade aged 8 to 10 years old.

Exclusion Criteria:

* medical history of heart disease, hypertension, diabetes, tuberculosis, asthma, hepatitis or nephritis;
* obesity caused by endocrine diseases or side effects of drugs;
* abnormal physical development like dwarfism or gigantism;
* physical deformity such as severe scoliosis, pectus carinatum, limp, obvious O-leg or X-leg;
* inability to participate in school sport activities;
* a loss in weight by vomiting or taking drugs during the past 3 months.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1627 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in body mass index (BMI） | 9months , 24 months and 36 months
  * weight and height will be combined to report BMI in kg/m^2
  * caculated by terminal value minus baseline value

SECONDARY OUTCOMES:
change in BMI z- score | 9months , 24 months and 36 months
  * measures of relative weight adjusted for child age and sex
  * caculated by terminal value minus baseline value
change in blood glucose | 9 months
  caculated by terminal value minus baseline value
change in blood lipids | 9 months
  * include TC, TG, LDL-C, HDL-C
  * caculated by terminal value minus baseline value
change in fasting insulin | 9 months
  caculated by terminal value minus baseline value
change in body fat percentage | 9 months
  caculated by terminal value minus baseline value
change in waist circumference | 9 months, 24 months and 36 months
  caculated by terminal value minus baseline value
change in weight | 9months, 24 months and 36 months
  caculated by terminal value minus baseline value
change in cardiorespiratory endurance test | 9 months, 24 months and 36 months
  caculated by terminal value minus baseline value

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, China

IPD SHARING:
Plan to Share IPD: No